CLINICAL TRIAL: NCT02967705
Title: Study on Pain Management Groups in Occupational Health Settings
Brief Title: Pain Management Groups in Occupational Health Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: Finnish Work Environment Fund (Other); Työterveys Helsinki (Helsinki city occupational health service) (Unknown)
Responsible Party: Principal Investigator, Helena Miranda, Project coordinator, Finnish Institute of Occupational Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 115395
Record Dates: First submitted 2016-10-20; First posted 2016-11-18 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Chronic Pain
Keywords: Pain Management; Chronic Pain; Health Services; Occupational Health
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain management group (Experimental): 6 + 1 meetings 2 hours each
  Interventions: Behavioral: Pain management group
- Treatment as usual (No Intervention): Waiting list - will receive treatment as usual

INTERVENTIONS:
Behavioral: Pain management group — Chronic pain patients participate in a peer group. They are provided information about chronic pain self-management based on biopsychosocial framework.
  Arms: Pain management group

SUMMARY:
This cluster randomized waiting-list controlled study will evaluate the effectiveness of pain management group activity organized by the OH on pain intensity and associated disability, and co-occurrence of mental or sleep problem in patients with chronic pain.

DETAILED DESCRIPTION:
Pain is very prevalent among the working population causing a considerable amount of work disability days. Pain management group therapy has shown to have a significant effect on chronic pain. However, little is known of the effect of such therapy on work disability. There are especially very few studies prescribing the effectiveness of pain management groups provided by the occupational health service.

ELIGIBILITY:
Inclusion Criteria:

- chronic pain + increased risk of work disability (based on a screening survey)

Exclusion Criteria:

* a malignant disease such as cancer, or severe mental illness such as depression causing significant functional disability.
* participating in another pain group elsewhere.
* in the middle of a major life crises such as divorce.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Change in pain intensity from before intervention to immediately after intervention and at 6 months
  self-reported questionnaire, 1-item question, scale 0-10, n=60
Pain self-efficacy | Change in pain self-efficacy from before intervention to immediately after intervention and at 6 months
  self-reported questionnaire, set of 10 questions, item response scale 0 - 6, n=60
Chronic pain acceptance | Change in chronic pain acceptance from before intervention to immediately after intervention and at 6 months
  self-reported questionnaire, set of 8 questions, item response scale 0 - 6, n=60
Fear-avoidance beliefs | Change in fear-avoidance beliefs from before intervention to immediately after intervention and at 6 months
  self-reported questionnaire, set of 3 questions, item response scale 0 - 6, n=18
Depressive symptoms | Change in depressive symptoms from before intervention to immediately after intervention and at 6 months
  self-reported questionnaire, 1-item question, response scale 0-10, n=60
Sleep problems | Change in sleep problems from before intervention to immediately after intervention and at 6 months
  self-reported questionnaire, 1-item question, response scale 0-10, n=60
Work ability | Change in work ability from before intervention to immediately after intervention and at 6 months
  self-reported questionnaire, 1-item question, response scale 0-10, n=60

SECONDARY OUTCOMES:
sickness absence | 6 months before and 6 months after intervention
  register based, number of sick leave days
health care contacts | 6 months before and 6 months after intervention
  register based, number of contacts to OHS

CONTACTS AND LOCATIONS:
Overall Officials: Helena Miranda, Dr.Med.Sc., Principal Investigator — Helsinki City OHS

IPD SHARING:
Plan to Share IPD: No